CLINICAL TRIAL: NCT03949933
Title: A Phase I Trial of Proton and Carbon Ion Radiation Dose Escalation in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Proton and Carbon Ion Radiotherapy for Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Guoliang Jiang, director of clinical technical committee, professor, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-PaCa2015-10
Record Dates: First submitted 2019-05-07; First posted 2019-05-14 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Pancreatic Carcinoma
Keywords: proton and carbon ion radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Protons; Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- proton and carbon ion radiotherapy (Experimental): proton and carbon ion radiotherapy
  Interventions: Radiation: proton and carbon ion radiotherapy

INTERVENTIONS:
Radiation: proton and carbon ion radiotherapy — proton and carbon ion radiotherapy

SUMMARY:
The aim of this study is to evaluate the toxicity and tolerance of proton and carbon ion radiotherapy (PCRT) for locally advanced pancreatic carcinoma (LAPC)

DETAILED DESCRIPTION:
The proton dose of 50.4GyE in 28 fractions was delivered to clinical target volume (CTV), and carbon ion as a boost dose to gross tumor volume (GTV) escalated from 12GyE to 18GyE with 3GyE per fraction in 3 dose levels. The dose limiting toxicity (DLT) was defined as CTCAE grade 3 or higher of non-hematological toxicity (G3). The acute and late toxicities, overall survival (OS), progression-free survival (PFS), local progression-free survival (LPFS) and distant metastasis-free survival (DMFS) were the endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. The histologically or cytologically confirmed, or the clinically diagnosed by clinical diagnosis criterion proposed by Pancreatic Cancer Committee of Chinese Anti-Cancer Association [15], which was based on evidences of (1). Typical symptoms of abdominal and/or back pain; (2). CA19-9 increased over the normal up limit; (3). A pancreatic mass shown on CT or MRI; and (4). SUV of PET-CT in mass increased compared to that in normal pancreas;
2. Unresectable LAPC defined by the criteria of (NCCN) guidelines (Version 1. 2013), or refusal to surgery;
3. Gastrointestinal tract (GI) not invaded;
4. ECOG Performance Status 0-1 within 30 days prior to registration;
5. Age of ≥ 18 years old;
6. Enough hematological function (white blood cell count ≥ 3.0×109/L; platelets ≥50×109/L; hemoglobin ≥ 90 g/L);
7. Enough liver and kidney functions (creatinine <110gmol/L; urea nitrogen <7.1mmol/L; bilirubin < 1.5 x ULN, ALT and AST ≤ 2.5 x ULN);
8. No evidence of distant metastases, based upon PET, CT, or MRI images of the chest, abdomen and pelvis within 30 days prior to registration;
9. Informed consent form obtained.

Exclusion Criteria:

1. No pathological evidence of malignant tumor;
2. ECOG>=2；
3. Liver, kidney and bone marrow function are poor and not adequate for treatment;
4. Side effect of previous treatment is not covered yet, eg. The interval between TACE and other anti-tumor therapy is less than one month;
5. Prior radiation therapy to the abdomen or radioactive particle implantation;
6. cardiac pacemaker or other metal implantation whose function may be disturbed by high energy beam or which affect the dose in target volume;
7. Dose constrain of normal liver, digested system and other OAR could not reach the expecting safe dose constrain;
8. The patient could not get benefit from proton or heavy ion radiotherapy in physician's opinion;
9. Comitant diseases or affecters which could affect the proton or heavy ion radiotherapy;
10. Pregnancy（blood or urine β-HCG certified）or lactation;
11. Drug or alcohol abused;
12. HIV positive, including received anti-retrovirus treatment; chronic hepatitis B virus replication stage; hepatitis C active stage; syphilis active stage;
13. HBV positive, hepatitis B virus replication stage, need to be treated with anti-virus treatment, but could not receive anti-virus treatment because of comitant disease;
14. Psychiatric history, possibly affecting the completion of treatment;
15. patients with serious complications that might affect radiotherapy， including 1）unstable angina pectoris requiring hospitalization in the last 6 months，congestive heart failure，myocardial infarction； 2）acute bacterial or systemic fungal infections； 3）exacerbation of chronic obstructive pulmonary disease ( COPD) or other respiratory system disease requiring hospitalization 4）hepatic function insufficiency or renal function insufficiency 5） immunosuppressed patients
16. patients with connective tissue disease such as active scleroderma or lupus and so on, which is contraindication for radiotherapy
17. patients can't understand treatment goal or unwilling/unable to sign up inform consent form；
18. no civil capability or limited civil capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Time interval from the start of radiotherapy to 3 months after the completion of radiotherapy
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
overall survival rate | 2 years
  overall survival rate
local progression-free survival | 2 years
  local progression-free survival
progression-free survivals | 2 years
  progression-free survivals

CONTACTS AND LOCATIONS:
Overall Officials: guoliang Jiang, Dr., Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No